CLINICAL TRIAL: NCT05167175
Title: A Single-center, Single-arm, Prospective Study to Investigate the Efficacy and Safety of Olaparib Combined With Abiraterone and Prednisone in mHSPC Patients With HRR Gene Mutation
Brief Title: The Study of Olaparib Combined With Abiraterone and Prednisone in mHSPC Patients With HRR Gene Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hongqian Guo (Other)
Collaborators: AstraZeneca (Industry); Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Hongqian Guo, Director of Urology Department, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROact
Record Dates: First submitted 2021-07-13; First posted 2021-12-22 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Prostate Carcinoma; Metastatic Prostate Cancer
Keywords: HRR; Olaparib; mCSPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention/Treatment (Experimental): Subjects will receive a regimen of Olaparib tablets 300 mg twice daily in combination with Abiraterone acetate 1000 mg plus Prednisone 5mg once daily until radiographic disease progression (assessed by the investigator according to RECIST1.1 and PCWG3) or intolerable adverse events (assessed by the investigator according to the actual clinical situation).
  Interventions: Drug: Olaparib tablet; Drug: Abiraterone acetate; Drug: Prednisone tablet

INTERVENTIONS:
Drug: Olaparib tablet — Lynparza (Olaparib tablets) 300 mg should be taken orally twice daily.
  Other Names: Lynparza
Drug: Abiraterone acetate — Qingkeshu (Abiraterone acetate tablets) 1000 mg should be taken orally once daily.
  Other Names: Qingkeshu
Drug: Prednisone tablet — Prednisone Tablets should be taken 5 mg once daily.

SUMMARY:
This is a single-center, single-arm, prospective study to assess the efficacy and safety of Olaparib combined with Abiraterone plus Prednisone in subjects with metastatic hormone sensitive prostate cancer (mHSPC) who carry deleterious germline or homologous recombination repair (HRR) mutations.

Olaparib is an oral, highly selective poly (ADP-ribose) polymerase (PARP) inhibitor that potently inhibits the activity of deoxyribonucleic acid repair polymerases. Abiraterone acetate (AA) is a prodrug of abiraterone that potently inhibits cytochrome P450c17, a key enzyme in androgen biosynthesis.

A total of 30 mHSPC subjects with HRR gene mutations that meet the criteria will be included in the study. Eligible subjects will receive oral Olaparib tablets 300 mg BID, combined with Abiraterone acetate 1000 mg QD plus Prednisone 5 mg, and the study will end when the primary endpoint radiographic progression-free survival (rPFS) data maturity reaches 60%. During the treatment and follow-up periods, all subjects will have regular visits to assess the efficacy and safety of Olaparib in combination with abiraterone acetate plus prednisone. Radiographic progression-free survival (rPFS), prostate-specific antigen response (PSA response rate), prostate-specific antigen progression-free survival (PSA-PFS), radiological objective response rate (ORR) and other indicators will be assessed and calculated.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects should fulfil the following criteria based on local regulations:

1. Provision of informed consent prior to any study specific procedures.
2. Adult male patients (age≥18 years old).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Histologically confirmed adenocarcinoma of the prostate.
5. Subjects must have at least 1 qualifying HRR gene mutation in tumor tissue by central lab (Glorious Med, shanghai, China).

   * Archival or new biopsies are acceptable.
   * Qualifying HRR gene mutations (deleterious or suspected deleterious gene alterations) are BRCA1, BRCA2, ATM, BARD1, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, RAD51B, RAD 51C, RAD51D and RAD54L mutations confirmed by the central lab.
6. The subject had a serum testosterone level ≤ 50 ng/dL (≤ 1.75 nmol/L) before enrollment.
7. Patients who have not undergone previous surgery must be taking and voluntarily continue taking LHRH analogues (agonists or antagonists) throughout the study treatment period.
8. Subjects must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Hemoglobin ≥ 10.0 g/dL without previous transfusion within 28 days.
   * Absolute neutrophil count ≥ 1.5 × 10^9/L.
   * Platelet count ≥ 100 × 10^9/L.
   * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN) specified.
   * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase) ≤ 2.5 × the specified ULN, unless liver metastases are present, in which case it must be ≤ 5 × ULN.
   * Estimated creatinine clearance ≥ 51 mL/min (estimated creatinine clearance = [140 - age (years)] × weight (kg)/(serum creatinine (mg/dL)×72)).
9. Male patients must use a condom during treatment and for 12 weeks after the last dose of Olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception ([see appendix C for acceptable methods]) if they are of childbearing potential
10. Subjects must have a life expectancy ≥ 16 weeks.
11. The subjects must volunteer and be capable of complying with the protocol for the duration of the study, including receiving treatment, attending scheduled visits and hospital examinations.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site) .
2. Previous enrolment in the present study.
3. Subjects participated in another clinical study with a drug or plan to participate in another interventional clinical study within 30 days prior to enrollment.
4. Prior treatment with any PARP inhibitor or any new hormone agent, including Olaparib, Niraparib, Abiraterone, Enzalutamide, Apalutamide, etc.
5. Prior chemotherapy with any DNA-damaging cytotoxic agent unless used to treat non-prostate cancer and the last dose was at least 5 years prior to enrollment in this study. For example: Patients previously treated with mitoxantrone or platinum-based chemotherapy for prostate cancer are excluded.
6. Patients who have received prior chemotherapy with any taxane. For example, patients who have received prior Docetaxel for prostate cancer are excluded.
7. Other malignancies within the last 5 years.
8. History of adrenal dysfunction.
9. Presence of persistent uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg). Subjects with a history of hypertension are allowed to participate if blood pressure could be controlled within these limits by antihypertensive therapy.
10. Uncontrolled or underlying cardiac disease on resting electrocardiogram (eg, but not limited to: unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QT prolongation > 500 ms with Fridericia correction, congenital long QT syndrome).
11. The subject had received any systemic anticancer therapy (except radiotherapy for palliative reasons) 3 weeks prior to study treatment.

    * Medications used to maintain castrate status are permitted as described in Inclusion Criteria 7. Drugs such as 5-α reductase inhibitors (finasteride, dutasteride), estrogen compounds and megestrol are considered as anticancer drugs and are prohibited at least 3 weeks before study treatment.
    * Treatment of bone metastases with denosumab or bisphosphonates such as zoledronic acid is allowed.
12. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, ritonavir, cobicistat, boceprevir or carbidetex-boosted protease inhibitors, indinavir, saquinavir, nelfinavir, baprevir, teicoplanavir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, sulfadiazine, fluconazole, diltiazem, vilapamil) requires a 2-week washout period prior to initiation of Olaparib therapy.
13. Concomitant use of strong CYP3A inducers (e.g. phenobarbital, empagliflozin, enzalutamide, phenytoin, rifampin, rifapentine, rifabutin, carbamazepine, nevirapine, and Forsythia leaf) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). If co-administered with phenobarbital or enzalutamide, a 5-week washout period is required before the start of Olaparib therapy and a 3-week washout period is required when co-administered with other drugs.
14. Subjects with major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
15. Subjects with previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
16. Long-term toxicity (CTCAE > grade 2) due to prior cancer therapy, excluding toxicity due to alopecia or use of LHRH agonists or antagonists.
17. Subjects with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML
18. Subjects with known brain metastases (confirmation of absence of brain metastases by scan is not required).
19. Subjects with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 4 weeks.
20. Subjects who are unable to swallow oral medication and/or have a gastrointestinal disorder that would interfere with absorption of the study drug.
21. Subjects with known allergic to Olaparib or Abiraterone acetate or any of the excipients of the two products.
22. Immunocompromised subjects, such as those with positive human immunodeficiency virus (HIV) serology.
23. Subjects with known active hepatitis (e.g. hepatitis B or C).
24. The subject has a serious, uncontrolled medical condition or non-malignant systemic disease, or an uncontrolled active infection. ( For example, but not limited to: uncontrolled arrhythmia, uncontrolled (with 12 weeks) myocardial infarction, unstable spinal cord compression, superior vena cava syndrome, uncontrolled seizures, extensive interstitial lung disease in both lungs, or psychiatric disease that would preclude informed consent.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | 18 month
  Time from the start of study drug to radiographic progression, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
PSA response rate | 18 month
  PSA response is defined as a ≥ 50% decline in PSA from baseline PSA value. This PSA decline must be confirmed as sustained by a second PSA value obtained ≥ 3 weeks later.
PSA Progression Free Survival (PSA-PFS) by Investigator | 18 month
  PSA-PFS is defined as the time from the start of study drug to the first PSA progression or death due to any cause without progression. PSA progression is defined as a first PSA increase greater than or equal to 25% of baseline and ≥ 2 ng/ml and confirmed a second time after 3 or more weeks.
Confirmed Objective Response Rate (ORR) by Investigator | 18 month
  ORR is the percentage of patients with at least one visit response of Complete response (CR) or Partial response (PR), in their soft tissue disease assessed by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), in the absence of progression on bone scan assessed by Prostate Cancer Working Group 3 (PCWG3)). Per RECIST v1.1, CR=Disappearance of all target lesions; PR = >=30% decrease in the sum of diameters of target lesions; For each treatment group, ORR is the number of patients with a CR and PR.

OTHER OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | 18 month
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No